CLINICAL TRIAL: NCT05636891
Title: Randomized, Double-blind, Parallel, Active Controlled Study to Compare Pharmacokinetic/Pharmacodynamic Parameters of Nanogen's Darbepoetin Alfa With Aranesp® (Amgen) in Treatment of Anemia in Chronic Kidney Disease Patients on Dialysis
Brief Title: Pharmacokinetic/Pharmacodynamic Parameters of NNG-DEPO (Stimus) With Aranesp® (Amgen) in Treatment of Anemia in CKD Patients on Dialysis
Acronym: CKD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Collaborators: Vietstar Biomedical Research (Industry); Clinical Research Consultants, Inc. (Industry); Clinical Research Viet Nam Skill Training And Consultant Company Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NNG06.1
Record Dates: First submitted 2022-10-13; First posted 2022-12-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease
Keywords: darbepoetin alfa; Nanogen; CKD; dialysis; treatment of anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimus (Experimental): Treatment: Nanogen's Darbepoetin alfa 10µg/0.4mL, 20µg/0.5mL, 40µg/0.4mL, 60µg/0.3mL, prefilled syringe
  Interventions: Biological: Stimus
- Aranesp (Active Comparator): Control: Amgen's Aranesp® 10µg/0.4mL, 20µg/0.5mL, 40µg/0.4mL, 60µg/0.3mL, prefilled syringe
  Interventions: Biological: Stimus

INTERVENTIONS:
Biological: Stimus — * NNG-DEPO (Darbepoetin alfa 10 mcg/0.4 mL, 20 mcg/0.5 mL, 40 mcg/0.4 mL, 60 mcg/0.3 mL) is available as a prefilled syringe in a sterile, colorless, glass tube.
  * Aranesp® (Darbepoetin alfa 10 mcg/ 0.4 mL, 20 mcg/ 0.5 mL, 40 mcg/ 0.4 mL, 60 mcg/ 0.3 mL) is manufactured by Amgen, as a pre-filled syringe in a sterile, glass tube, colourless.
  Storage: 2-8ºC, not frozen. The process of transporting and storing the drug must ensure the temperature in the range of 2-8ºC.
  NNG-DEPO/Aranesp is administered subcutaneously (or intravenously for patients with PK-PD in the previous IV group), at a dose of 0.75 g/kg initially, every 2 weeks at the second visit.
  IPs will be prepared according to standard procedure (SOP). Dosage adjustment guideline:
  Patients will have hemoglobin levels monitored every 2 weeks. The investigators will evaluate and adjust the dose of Darbepoetin alfa to maintain the Hb levels within the target range (10 - 12 g/dL)

SUMMARY:
This is a double-blind, randomized, active-control study with 2-study arms-darbepoetin alfa biosimilar and Aranesp, noninferiority trial design in dialysis patients. Dialysis patients will be randomized into 1:1 ratio to receive either Darbepoetin alfa or Aranesp 0.75 µg/kg by subcutaneous injection every other week for 24 weeks.

Pharmacokinetic/pharmacodynamic parameters for evaluation are assessed as per study endpoints at defined time points on all patients.

During the treatment, dose adjustments will be made as necessary to achieve a hemoglobin response, defined as maintaining Hb in target range 10 - 12 g/dL.

DETAILED DESCRIPTION:
PHASE OF TRIAL: I SAMPLE SIZE: 43 for pharmacokinetic/pharmacodynamic parameters TARGET POPULATION: Patients with chronic kidney disease undergoing dialysis

STUDY GROUPS:

1. Darbepoetin alfa (Nanogen) SC 0.75 µg/kg Q2W, for 24 weeks.
2. Aranesp® (Amgen) SC 0.75 µg/kg Q2W, for 24 weeks.

PK ASSESSMENT: Blood samples for PK assessments will be collected at:

* IV: time zero (predose) before injection of study drug and then after 0.25, 0.5, 4, 12, 24, 48, 96, 144, 240 and 336 hours post-dose.
* SC: time zero (predose) before injection of study drug and then after 4, 12, 24, 48, 96, 144, 240 and 336 hours post-dose.

PD ASSESSMENT: Blood samples for PD assessments will be collected at time zero (predose) before injection of study drug and then after 24, 48, 96, 144, 240 and 336 hours post-dose.

SAFETY AND TOLERABILITY ASSESSMENT:

Safety and tolerability assessments will be performed at each visit. Following variables will be considered to define the safety and tolerability of investigational drugs:

* Clinical adverse events (AEs): frequency of AEs, overall and by intensity.
* Severe clinical adverse events (SAEs): frequency of AEs, overall and by intensity.
* Symptoms directed physical examination including body weight, and vital signs during treatment period: mean change from baseline and the frequency of clinically relevant changes from baseline.
* Laboratory tests: frequency of clinically relevant changes from baseline.
* The frequency of any concomitant medication administered to treat any adverse events.
* Presence of anti-bodies to darbepoetin alfa (immunogenicity).

ELIGIBILITY:
Inclusion Criteria

* The patients signed the informe consent form and adhere to study visit schedule.
* Male or female patients aged from 18 to 65 years.
* Patients on hemodialysis or peritoneal dialysis for at least 3 months and have Hb baseline <10 g/dL during the screening period.
* Have transferrin saturation ≥ 20%, serum ferritin ≥ 200 ng/mL, vitamin B12 and folate within the normal range.
* Have expected survival of at least 6 months from time of enrollment (by investigator's assessment).
* Women childbearing age must agree to use medically acceptable methods of contraception during the study and for 6 months after the last study treatment.
* The patient does not have any serious medical conditions that may affect to study treatment compliance.

Exclusion Criteria

* Uncontrolled hypertension over 2 weeks prior to and within the screening period (BP ≥ 160/90 mmHg).
* Patients treated with Darbepoetin alfa or r-HuEPO within 4 weeks prior to enrollment.
* Patients with Uncontrolled diabetes mellitus with HbA1C ≥ 10%.
* Congestive Heart Failure of grade 3 or 4 as New York Heart Association classification.
* History of unstable angina or myocardial infarction within 6 months.
* History of Grand mal seizures in last 2 years.
* Present with severe hyperparathyroidism (iPTH >1500 pg/mL for Dialysis).
* History of major surgery within 12 weeks prior to screening.
* Systemic hematologic disorders including sickle cell anemia, myelodysplastic syndromes, hematological malignancy, myeloma and hemolytic anemia.
* Systemic infections, active inflammatory diseases and malignancies.
* Active liver disease or hepatic with liver enzymes AST and ALT raised > 2-times of laboratory normal values, child B or child C cirrhosis.
* Are being treated with androgen therapy within the 8 weeks prior to the screening period.
* Pregnant or suspected pregnant women, breast-feeding women.
* Patients scheduled for any transplant procedure within 6 months of screening or with a previous history of kidney transplantation.
* Patients who are hypersensitive to any of substances of investigational product.
* Patients using drugs that can affect the concentration of Hb in the blood (except blood-forming drugs such as iron, folic acid).
* Patients with seropositivity to HIV, HBV or anti-HCV.
* Patients having acute tuberculosis or any acute bacterial infection within 1 month prior to the screening.
* Patient has occult blood in stool or any other known source of internal bleeding and confirmed gastrointestinal bleeding by endoscopy.
* Patients with blood transfusion due to acute bleeding within 12 weeks prior to screening period.
* Patients with a history of immunosuppressive therapy within 1 month.
* The patient is suffering from advanced cancer.
* Patients having participated in any other clinical trial within 1 month prior to the screening period.
* The patient had any medical condition that the investigator assessed as affecting the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-09-19 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
PK parameters comparison between NNG-DEPO and Aranesp®: Cmax | IV:Assessed predose and at 0.25; 0.5; 4;12;24;48;96;144;240;336 hours postdose/ SC: Assessed predose and at 4;12;24;48;96;144;240;336 hours postdose
  Serum peak concentrations (Cmax)
PK parameters comparison between NNG-DEPO and Aranesp®: AUC(0, t) | IV:Assessed predose and at 0.25; 0.5; 4;12;24;48;96;144;240;336 hours postdose/ SC: Assessed predose and at 4;12;24;48;96;144;240;336 hours postdose
  Area under the curve from 0 to t (AUC 0-t)

SECONDARY OUTCOMES:
PD parameters comparison between NNG-DEPO and Aranesp®: Cmax of reticulocytes | Assessed predose and at and at 24;48;96;144;240;336 hours postdose
  Serum peak concentrations (Cmax) of reticulocytes
PD parameters comparison between NNG-DEPO and Aranesp®: AUC(0, t) of reticulocytes | Assessed predose and at and at 24;48;96;144;240;336 hours postdose
  Area under the curve from 0 to t (AUC 0-t) of reticulocytes
PD parameters comparison between NNG-DEPO and Aranesp®: Tmax of reticulocytes | Assessed predose and at and at 24;48;96;144;240;336 hours postdose
  Time for the drug to reach peak concentration (Tmax) of reticulocytes
PK parameters comparison between NNG-DEPO and Aranesp®:Tmax | IV:Assessed predose and at 0.25; 0.5; 4;12;24;48;96;144;240;336 hours postdose/ SC: Assessed predose and at 4;12;24;48;96;144;240;336 hours postdose
  Time for the drug to reach peak concentration (Tmax)
PK parameters comparison between NNG-DEPO and Aranesp®: AUC(0,∞) | IV:Assessed predose and at 0.25; 0.5; 4;12;24;48;96;144;240;336 hours postdose/ SC: Assessed predose and at 4;12;24;48;96;144;240;336 hours postdose
  Area under the curve from 0 to ∞ (AUC0-∞)
PK parameters comparison between NNG-DEPO and Aranesp®:T1/2 | IV:Assessed predose and at 0.25; 0.5; 4;12;24;48;96;144;240;336 hours postdose/ SC: Assessed predose and at 4;12;24;48;96;144;240;336 hours postdose
  Half-life (T1/2)
PK parameters comparison between NNG-DEPO and Aranesp®: CL/F | IV:Assessed predose and at 0.25; 0.5; 4;12;24;48;96;144;240;336 hours postdose/ SC: Assessed predose and at 4;12;24;48;96;144;240;336 hours postdose
  CL/F
PK parameters comparison between NNG-DEPO and Aranesp®:Vz/F | IV:Assessed predose and at 0.25; 0.5; 4;12;24;48;96;144;240;336 hours postdose/ SC: Assessed predose and at 4;12;24;48;96;144;240;336 hours postdose
  Vz/F
PK parameters comparison between NNG-DEPO and Aranesp®: λz. | IV:Assessed predose and at 0.25; 0.5; 4;12;24;48;96;144;240;336 hours postdose/ SC: Assessed predose and at 4;12;24;48;96;144;240;336 hours postdose
  λz.
Proportion of the adverse events (AE) including physical examinations, vital signs, and clinical laboratory investigations. | Week 0 (Assessed predose)- Week 24]
  Rate of AE and SAE occurence

CONTACTS AND LOCATIONS:
Locations (1):
- NANOGEN Pharmaceutical Biotechnology JSC, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided